CLINICAL TRIAL: NCT01078753
Title: A Double-blind, Placebo-controlled, Phase III Comparative Study With FE992026 in Children and Adolescents With Reduced Night-time Urinary Osmolarity-type Nocturnal Enuresis
Brief Title: Study With Two Different Doses of Desmopressin Orally Lyophilisate Tablet With Nocturnal Enuresis
Acronym: PNE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FE992026 CS35
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-09

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desmopressin (Experimental): During treatment period I participants received 120 μg per day desmopressin oral lyophilisate tablet for 14 days. Participants for whom treatment was effective (a reduction of ≥ 75% from Baseline in the number of wet nights), and who showed no problems with tolerability, continued to receive the same treatment for a further 14 days in treatment period II. Participants for whom efficacy was inadequate (a reduction of <75% from Baseline in the number of wet nights), but who showed no tolerability problems, received an increased dose of desmopressin oral lyophilisate tablet 240 µg for 14 days in treatment period II.
  Interventions: Drug: Desmopressin
- Placebo (Placebo Comparator): Participants received matching placebo tablets during treatment periods I and II according to the same efficacy criteria as participants in the Desmopressin treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin — Desmopressin oral lyophilisate tablet, 120 μg or 240 μg, administered sublingually once a day 1½ hours before bedtime.
  Other Names: FE992026; desmopressin melt; Minirin
  Arms: Desmopressin
Drug: Placebo — Placebo oral lyophilisate tablet was administered sublingually once a day 1½ hours before bedtime.
  Arms: Placebo

SUMMARY:
This is multi-center, randomized, placebo-controlled, parallel-group, double-blind, dose-escalating clinical trial designed to assess the efficacy and safety of desmopressin orally lyophilisate for the treatment of nocturnal enuresis "with decreased nighttime urinary osmolality."

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed nocturnal enuresis with reduced nighttime urinary osmolality
* Age 6 or above but under 16 regardless of gender
* Out-patient
* Had 10 or more wet nights during the 14-day baseline period and at least 4 wet nights in each respective week
* Deemed healthy by the investigator
* Able to agree to and comply with fluid-intake restriction during the clinical trial and matters specified in the clinical trial protocol
* Consent from the pediatric patient's legally acceptable representative
* Demonstrate an understanding about this clinical trial after receiving an explanation corresponding to the prospective subject's intelligibility
* Show no possibility of being a nursing mother or pregnant, or becoming pregnant
* If under drug or medical therapy other than Desmopressin for treating nocturnal enuresis: able to discontinue such treatment

Exclusion Criteria:

* Suffer from enuresis with an underlying disease
* Participated in another clinical trial within six months preceding consent
* Used an intranasal Desmopressin in the past
* Presently undergoing a systemic antibiotic treatment, a treatment with an antidiuretic or a drug that affects urinary concentration, or a drug or medical therapy for overactive bladder
* Have an anomaly or a disease that may affect the oral absorption of drug products
* Hard to get cooperation from subject by school refusal, punishment or bullying
* Deemed by the investigator to be inappropriate to participate in this trial
* Unable to be placed on water-intake restriction starting from two hours before bedtime
* Evidence of hepatic, renal, cardiac, or pulmonary dysfunction

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (15):
- Japan (15):
  - Akita University Hospital, Akita, Akita
  - Hiroshima Red Cross Hospital and Atomic Bomb Survivors Hospital, Hiroshima, Hiroshima
  - Showa Hospital, Amagasaki, Hyōgo
  - Shinko-Kakogawa Hospital, Kakogawa, Hyōgo
  - Tamura Children's Clinic, Mito, Ibaraki
  - Shinbo Child Clinic, Yokohama, Kanagawa
  - Aikawa Station Clinic, Niigata, Niigata
  - Kansai Medical University Hirakata Hospital, Hirakata, Osaka
  - Kitano Hospital, Osaka, Osaka
  - Saitama Childrens Medical Centre, Saitama, Saitama
  - Shintoshin Child Clinic, Saitama, Saitama
  - Takesue Children's Clinic, Musashino, Tokyo
  - Juntendo University Nerima Hospital, Nerima City, Tokyo
  - Saitoh Pediatric Medical Clinic, Nishitōkyō, Tokyo
  - Hoashi Children's Psychological Clinic, Setagaya City, Tokyo

REFERENCES:
- [Derived] Hahn D, Stewart F, Raman G. Desmopressin for nocturnal enuresis in children. Cochrane Database Syst Rev. 2025 Jul 29;7(7):CD002112. doi: 10.1002/14651858.CD002112.pub2. PMID 40728007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 174 subjects consented and entered the 14-day screening period during which Baseline characteristics regarding enuretic episodes were established. Eligible patients who met the criterion were randomized 1:1 to receive either desmopressin or matching placebo.
  Randomization was stratified by gender, age and number of wet nights at Baseline.
Period: Treatment Period I
Arm/Group | Desmopressin | Placebo
Started | 45 | 44
Full Analysis Set | 44 (One patient was excluded from the full analysis set due to failure to satisfy the entry criteria.) | 44
Completed | 45 | 44
Not Completed | 0 | 0
Period: Treatment Period II
Arm/Group | Desmopressin | Placebo
Started | 45 (Desmopressin 120 µg - 4 participants Desmopressin 240 µg - 41 participants) | 44
Full Analysis Set | 44 (One patient was excluded from the full analysis set due to failure to satisfy the entry criteria.) | 44
Completed | 45 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desmopressin | Placebo | Total
Number analyzed (Participants) | 45 | 44 | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 8.2 (1.6) | 8.1 (1.4) | 8.1 (1.5)
Age, Customized [Number; unit: participants]
  6 to 9 years old | 36 | 36 | 72
  10 to15 years old | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 28 | 23 | 51
Region of Enrollment [Number; unit: participants]
  Japan | 45 | 44 | 89
Height [Mean (Standard Deviation); unit: cm] | 128.14 (11.30) | 127.68 (8.61) | 127.92 (10.01)
Weight [Mean (Standard Deviation); unit: kg] | 27.59 (8.40) | 27.01 (5.32) | 27.30 (7.01)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m˄2] | 16.46 (2.47) | 16.43 (1.77) | 16.44 (2.14)
Number of Wet Nights during Baseline [Mean (Standard Deviation); unit: days] — Number of Wet Nights recorded during the 14-day Baseline period.
  days | 12.2 (1.5) | 12.4 (1.5) | 12.3 (1.5)
Number of Wet Nights during Baseline by stratification criteria [Number; unit: participants] — The number of wet nights recorded during the 14-day Baseline period is reported for each of the stratification categories.
  participants
    10 to 13 wet nights | 32 | 30 | 62
    14 wet nights | 13 | 14 | 27
Prior treatment of Nocturnal Enuresis with Drugs [Number; unit: participants]
  No prior treatment | 45 | 44 | 89
  Prior treatment received | 0 | 0 | 0
Prior treatment of Nocturnal Enuresis with Therapy [Number; unit: participants] — Therapies for treatment of Nocturnal Enuresis might include life-skill guidance, bladder control training, psychotherapy, or behaviour conditioning therapy.
  participants
    No prior therapy | 0 | 0 | 0
    Prior therapy | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Wet Nights Between Baseline and Treatment Period II
Description: The number of wet nights was recorded by participants (or their caregivers) in a daily diary. The difference was calculated from the number of wet nights during the 14-day Baseline Period minus the number of wet nights during the 14-day Treatment Period II.
Time Frame: Baseline (14-day period prior to starting study treatment) and Treatment Period II (weeks 3-4 after treatment initiation).
Population: The Full Analysis Set (FAS) included all participants who received at least one dose of study treatment, satisfied all the major eligibility criteria and for whom efficacy data was obtained.
Measure: Least Squares Mean (95% Confidence Interval); unit: wet nights
Arm/Group | Desmopressin | Placebo
Number analyzed (Participants) | 44 | 44
wet nights | 3.264 [2.126 to 4.402] | 1.451 [0.333 to 2.570]
Statistical Analysis 1: Comparison: Desmopressin vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA — Desmopressin was considered to be superior to Placebo if the p-value for the comparison was < 0.05 and the reduction from Baseline in number of wet nights was larger in the FE992026 group than in the Placebo group; Factors in the analysis were Gender (male, female), age (6≤x≤9, 10≤x≤15), number of wet nights at Baseline (10≤x≤13, x=14), and treatment group; Least Squares Mean Difference = 1.813, 95% CI 2-sided [0.462 to 3.163]

2. Secondary Outcome: Change in Number of Wet Nights Between Baseline and Treatment Period I
Description: The number of wet nights was recorded by participants (or their caregivers) in a daily diary. The difference was calculated from the number of wet nights during the 14-day Baseline Period minus the number of wet nights during the 14-day Treatment Period I.
Time Frame: Baseline (14-day period prior to starting study treatment) and Treatment Period I (weeks 1-2 after treatment initiation).
Population: The Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: wet nights
Arm/Group | Desmopressin | Placebo
Number analyzed (Participants) | 44 | 44
wet nights | 2.946 [1.815 to 4.078] | 1.317 [0.205 to 2.428]
Statistical Analysis 1: Comparison: Desmopressin vs Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares mean Difference = 1.629, 95% CI 2-sided [0.287 to 2.972]

3. Secondary Outcome: Change in Number of Wet Nights Between Treatment Periods I and II
Description: The number of wet nights was recorded by participants (or their caregivers) in a daily diary. The difference was calculated from the number of wet nights during the 14-day Treatment Period I minus the number of wet nights during the 14-day Treatment Period II.
Time Frame: Treatment Period I (weeks 1-2) and Treatment Period II (weeks 3-4)
Population: The full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: wet nights
Arm/Group | Desmopressin | Placebo
Number analyzed (Participants) | 44 | 44
wet nights | 0.318 [-0.653 to 1.289] | 0.135 [-0.819 to 1.088]
Statistical Analysis 1: Comparison: Desmopressin vs Placebo; Test type: Superiority or Other; p = 0.752, ANCOVA; Factors in the analysis included Gender (male, female), age (6≤x≤9, 10≤x≤15), number of wet nights at Baseline (10≤x≤13, x=14), and treatment group; Least Squares Mean Difference = 0.183, 95% CI 2-sided [-0.968 to 1.335]

ADVERSE EVENTS:
Time Frame: 4 weeks (periods I + II)
Arm/Group | Desmopressin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 18/45 | 14/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Desmopressin (N=45) | Placebo (N=44)
Empyema (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 6
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin papilloma (Skin and subcutaneous tissue disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Feeling hot (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Blood calcium decreased (Investigations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention